CLINICAL TRIAL: NCT07103252
Title: BOOST- Blood Flow Restriction Therapy to Optimize Muscle Size and Strength in Recovery From Lower Limb Orthopaedic Trauma
Brief Title: Blood Flow Restriction Therapy to Optimize Muscle Size and Strength in Recovery From Lower Limb Fractures
Acronym: BOOST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: AO North America (Other)
Responsible Party: Principal Investigator, Kelly A. Lefaivre, MD, MSc, FRCSC, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H25-01080
Record Dates: First submitted 2025-07-25; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Tibial Fracture
Keywords: Blood Flow Restriction Therapy; Lower Extremity; Tibia; Feasibility Study; Leg Injuries; Fractures, Bone; Quadriceps Muscle
MeSH Terms: conditions — Tibial Fractures; Leg Injuries; Fractures, Bone | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the treatment arm or control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Physiotherapy without BFRT
- Blood Flow Restriction Therapy (BFRT) (Experimental): Physiotherapy with BFRT
  Interventions: Other: Blood Flow Restriction Therapy

INTERVENTIONS:
Other: Blood Flow Restriction Therapy — Personalized Blood Flow Restriction Therapy uses an an inflatable cuff (Delfi PTS system) around the upper thigh which partially restricts arterial inflow during exercise. BFR allows for similar improvements of muscular strength and muscle mass as traditional heavy load strength training while using significantly lower loads. The reduced stress on supporting tissues ( tendons, joints, bones and ligaments) allows people who normally couldn't tolerate high loads to enhance their strength and muscle mass.
  Arms: Blood Flow Restriction Therapy (BFRT)

SUMMARY:
This study will assess the feasibility and effectiveness of blood flow restriction therapy in patients with tibia fractures (or lower leg bone). Personalized blood flow restriction therapy has shown to help people regain muscle size and strength after surgical treatment by allowing them to be able to start physiotherapy on their injured leg sooner. This study aims to evaluate the feasibility and effectiveness of personalized blood flow restriction therapy to improve thigh muscle size and strength in patients with lower limb tibia fractures which require a period of non-weightbearing.

DETAILED DESCRIPTION:
Lower limb fractures constitute the largest burden of fracture care globally. It is well documented that major upper and lower extremity trauma results in significant disability, with a protracted trajectory of recovery. A large proportion of these fracture can require a period of immobilization or protected weight bearing for up to 12 weeks depending on the nature, location and treatment of the fracture. Loss of muscle bulk and functional strength can occur with immobilization and disuse in as early as five days, and is confounded by severity of injury. Rehabilitation of these patients is focused on regaining range of motion, muscle strength and return to function. Traditional regimens to increase muscle size require exercises to be performed at high loads and intensities, typically at 60%-70% of a person's one repetition maximum. Due to the prolonged period of weight bearing protection and/or immobilization, and the recovery from the traumatic injury itself, most patients are unable to engage in high intensity and load exercises. This limits their ability to improve muscle size and strength and in turn slows down their return to function.

Blood flow restriction therapy (BFRT) originated in the 1960s in Japan. However, this initial approach was wrought with poor safety and reliability. The implementation of the automatic pneumatic tourniquet in 1979 allowed for the pressure applied by the tourniquet to be reliably controlled and replicated. Since then, multiple studies have been done to improve upon the technique, with the main aims to identify the optimal occlusion pressure and extent of blood flow restriction.

Blood flow restriction works on the principle of restricting arterial inflow and occluding venous outflow from the chosen limb. The personalized aspect is drawn from the fact that the pressure applied is a pre-determined percentage of the patient's Limb Occlusion Pressure (LOP). LOP is defined as the minimum pressure required, at a specific time by a specific tourniquet cuff applied to a specific patient's limb at a specific location, to stop the flow of arterial blood into the limb distal to the cuff. Benefits have been shown with blood flow restriction at 40%-80% of the patient's LOP. Further, despite the relationship between blood flow and fracture healing, studies in upper limb fractures have demonstrated that the reduced blood flow does not have a detrimental effect on bony union.

Personalized blood flow restriction therapy (BFRT) can help achieve similar muscle growth by performing exercises at lower loads and intensities (20%-30%) of one repetition maximum. There is significant excitement around this concept in elective orthopaedics, and this treatment modality has been shown to be effective in rehabilitation from ACL reconstruction, total knee replacements, wrist fractures and Achilles tendon ruptures. Although what is known about recovery and long-term disability in lower extremity orthopaedic trauma patients makes them an obvious candidate for this, there is a lack of evidence for use in lower limb fractures. With this pilot study, the investigators hope to demonstrate the feasibility of conducting a larger RCT on this topic.

Hypotheses The investigators hypothesize that personalized BFRT will be tolerated by patients from 2 weeks post injury with increasing tolerance overtime. Personalized BFRT will demonstrate an increase in quadriceps muscle size and strength in the injured leg at 12 weeks following injury. The treatment effects of BFRT on lower extremity strength at 12 weeks in fracture patients will be used to inform the sample size calculation of a future definitive trial. The investigators further hypothesize that the proposed pilot trial will demonstrate feasibility of a future definitive trial.

Research design and methods This is a pilot study at a Level 1 Trauma Center (Vancouver General Hospital) involving patients with a peri-articular tibial fracture (treated operatively or non-operatively) which require a minimum 6 weeks of protected weight bearing (non weight bearing or partial weight bearing). Patients will be randomised to one of two groups - Physiotherapy with or without Blood Flow Restriction Therapy (PT with BFRT or PT without BFRT). Potential patients will be identified in the Orthopaedic Trauma outpatient clinic and physiotherapy departments. Recruitment and screening will be carried out as approved by the UBC Clinical Research Ethics Board. All patients presenting with a peri-articular tibial fracture (treated operatively or non-operatively) will be pre-screened, assigned a screening number, and recorded in a de-identified site screening log by the Orthopaedic Trauma research team. Those deemed potentially eligible will be approached by the research personnel. Informed, voluntary consent will be obtained from patients in a non-coercive manner. Patients will be enrolled for biweekly physiotherapy treatments from week 2 to week 12 post injury or post surgery. They will remain non-weightbearing for 6 weeks following the injury or surgery (first 4 weeks of physiotherapy). They Both groups will have standard clinical follow up at 2 weeks, 6 weeks and 12 weeks post injury/surgery.

Once local ethics approval and the pneumatic tourniquet have been received and the pneumatic tourniquet, the training planned for two of our hospital physiotherapists will be finalized. These therapists work full time in the outpatient setting, which is dedicated to the care of injured patients, and where baseline therapy is completely funded by the local Health Authority. Local expertise for training, and preliminary collaborations have been established. Patients will be assigned to one of two of these physiotherapists regardless of whether they are allocated to the PT with BFRT or PT without BFRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19-60 who have sustained an isolated (single bone/area as per AO/OTA classification) unilateral lower limb fracture of the tibia that requires a period of 6 weeks of protected weight bearing (non-weight bearing or toe touch weight bearing)
2. Must speak English
3. Must be able to comply with protected weight bearing instructions for at least 6 weeks
4. Must be able to consent for inclusion into the trial

Exclusion Criteria:

1. Patients who have sustained multiple fractures in the same limb (i.e. AO/OTA 3 and 4, or 4 and 8 etc).
2. Patients who have a neurovascular injury associated with the fracture
3. Patients who have sustained bilateral lower limb injuries
4. Patients aged <19 and >60
5. Patients with known peripheral vascular disease or vascular repair
6. Patients with known coagulation disorders
7. Patients with compartment syndrome
8. Patients with free tissue transfer for soft tissue coverage
9. Patients with ongoing VTE or infection in the affected limb
10. Non-ambulatory patients
11. Patients who are pregnant

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants who consent to participate | 12 weeks
  Percentage of participants approached for recruitment who consent to study participation
Number of participants self-reporting adherence to treatment protocol | 12 weeks
  Percentage of participants enrolled in the study who report to completing their prescribed post injury physiotherapy sessions
Number of participants missing data on regular assessment | 12 weeks
  Percentage of participants with missing data on regular assessment
Number of participants who withdraw from the study | 12 weeks
  Percentage of participants enrolled in the study who withdraw before completion of the study
Number of participants who complete follow up at 12 weeks | 12 weeks
  Percentage of enrolled participants who complete all follow up visits
Muscle strength tension and compression in pounds | 0, 2, 6, 12 weeks post injury/surgery
  Muscle strength of participants measured as force, tension and compression in pounds, in the affected limb using a dynamometer force gauge (ergoFET Digital Force Gauge)
Muscle size of the affected limb measured in centimeters | 0, 2, 6, 12 weeks post injury/surgery
  Muscle size of participants estimated by measuring muscle circumference of thigh at 10 cm above superior pole of patella in affected limb
Range of motion in degrees | 0, 2, 6, 12 weeks post injury/surgery
  Range of motion (degrees) of participants' knees (flexion, extension and rotation) and ankles (dorsiflexion and plantar flexion) using a goniometer.
Physical and mental health (SF12) | 0, 2, 6, 12 weeks post injury/surgery
  Physical and mental health of participants assessed using the short form health survey (SF12)
Ambulatory status | 0, 2, 6 and 12 weeks post the injury/surgery
  Percentage of participants who do or do not require a walking aid including cane, walker, wheelchair, or other.

OTHER OUTCOMES:
Limb Occlusion Pressure (LOP) in millimeters of mercury (mmHg) | 0, 2, 6, 12 weeks post injury/surgery
  Participants' maximum percentage of Limb Occlusion Pressure (LOP) in millimeters of mercury (mmHg) at which all exercises could be completed
Number of participants with incomplete Limb Occlusion Pressure (LOP) | 0, 2, 6, 12 weeks post injury/surgery
  Number of participants who could not complete the exercises at any percentage of Limb Occlusion Pressure (LOP)

CONTACTS AND LOCATIONS:
Overall Officials: David Stockton, MD MSc FRCSC, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
1. Will Individual participant data be available? Yes- only as permitted by UBC's Clinical Research Ethics Board
  2. What data: Individual participant data that underlie the results reported in an published article, after deidentification (text, tables, figures) only as permitted by UBC's Clinical Research Ethics Board
  3. Other documentation: Study protocol, statistical analysis plan, informed consent
  4. When data is available: Beginning 3 months and ending 24 months following publication.
  5. With whom: Researchers whose proposed use of the data has been approved by UBC's Clinical Research Ethics Board.
  6. Types of analyses: To achieve the aims in the proposal approved by UBC's Clinical Research Ethics Board.
  7. Data made available: proposals may be submitted up to 24 months following article publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 24 months following publication.
Access Criteria: Individual participant data that underlie the results reported in a published article, after deidentification (text, tables, figures) only as permitted by UBC's Clinical Research Ethics Board. Researchers whose proposed use of the data has been approved by UBC's Clinical Research Ethics Board.

REFERENCES:
- [Background] Avery KN, Williamson PR, Gamble C, O'Connell Francischetto E, Metcalfe C, Davidson P, Williams H, Blazeby JM; members of the Internal Pilot Trials Workshop supported by the Hubs for Trials Methodology Research. Informing efficient randomised controlled trials: exploration of challenges in developing progression criteria for internal pilot studies. BMJ Open. 2017 Feb 17;7(2):e013537. doi: 10.1136/bmjopen-2016-013537. PMID 28213598
- [Background] Franz A, Ji S, Bittersohl B, Zilkens C, Behringer M. Impact of a Six-Week Prehabilitation With Blood-Flow Restriction Training on Pre- and Postoperative Skeletal Muscle Mass and Strength in Patients Receiving Primary Total Knee Arthroplasty. Front Physiol. 2022 Jun 14;13:881484. doi: 10.3389/fphys.2022.881484. eCollection 2022. PMID 35774280
- [Background] Hughes L, Rosenblatt B, Haddad F, Gissane C, McCarthy D, Clarke T, Ferris G, Dawes J, Paton B, Patterson SD. Comparing the Effectiveness of Blood Flow Restriction and Traditional Heavy Load Resistance Training in the Post-Surgery Rehabilitation of Anterior Cruciate Ligament Reconstruction Patients: A UK National Health Service Randomised Controlled Trial. Sports Med. 2019 Nov;49(11):1787-1805. doi: 10.1007/s40279-019-01137-2. PMID 31301034
- [Background] Centner C, Lauber B, Seynnes OR, Jerger S, Sohnius T, Gollhofer A, Konig D. Low-load blood flow restriction training induces similar morphological and mechanical Achilles tendon adaptations compared with high-load resistance training. J Appl Physiol (1985). 2019 Dec 1;127(6):1660-1667. doi: 10.1152/japplphysiol.00602.2019. Epub 2019 Nov 14. PMID 31725362
- [Background] Fan Y, Bai D, Cheng C, Tian G. The effectiveness and safety of blood flow restriction training for the post-operation treatment of distal radius fracture. Ann Med. 2023;55(2):2240329. doi: 10.1080/07853890.2023.2240329. PMID 37505919
- [Background] Lixandrao ME, Ugrinowitsch C, Laurentino G, Libardi CA, Aihara AY, Cardoso FN, Tricoli V, Roschel H. Effects of exercise intensity and occlusion pressure after 12 weeks of resistance training with blood-flow restriction. Eur J Appl Physiol. 2015 Dec;115(12):2471-80. doi: 10.1007/s00421-015-3253-2. Epub 2015 Sep 1. PMID 26323350
- [Background] Noordin S, McEwen JA, Kragh JF Jr, Eisen A, Masri BA. Surgical tourniquets in orthopaedics. J Bone Joint Surg Am. 2009 Dec;91(12):2958-67. doi: 10.2106/JBJS.I.00634. PMID 19952261
- [Background] Spranger MD, Krishnan AC, Levy PD, O'Leary DS, Smith SA. Blood flow restriction training and the exercise pressor reflex: a call for concern. Am J Physiol Heart Circ Physiol. 2015 Nov;309(9):H1440-52. doi: 10.1152/ajpheart.00208.2015. Epub 2015 Sep 4. PMID 26342064
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Larose G, Roffey DM, Broekhuyse HM, Guy P, O'Brien P, Lefaivre KA. Trajectory of Recovery following ORIF for Distal Radius Fractures. J Wrist Surg. 2023 Jul 13;13(3):230-235. doi: 10.1055/s-0043-1771045. eCollection 2024 Jun. PMID 38808181
- [Background] Middleton SD, Guy P, Roffey DM, Broekhuyse HM, O'Brien PJ, Lefaivre KA. Long-Term Trajectory of Recovery Following Pilon Fracture Fixation. J Orthop Trauma. 2022 Jun 1;36(6):e250-e254. doi: 10.1097/BOT.0000000000002312. PMID 34799544
- [Background] GBD 2019 Fracture Collaborators. Global, regional, and national burden of bone fractures in 204 countries and territories, 1990-2019: a systematic analysis from the Global Burden of Disease Study 2019. Lancet Healthy Longev. 2021 Sep;2(9):e580-e592. doi: 10.1016/S2666-7568(21)00172-0. PMID 34723233